CLINICAL TRIAL: NCT02954653
Title: A PHASE 1 DOSE ESCALATION STUDY TO EVALUATE THE SAFETY, PHARMACOKINETICS AND PHARMACODYNAMICS OF INTRAVENOUS PF-06747143, ADMINISTERED AS SINGLE AGENT OR IN COMBINATION WITH STANDARD CHEMOTHERAPY IN ADULT PATIENTS WITH ACUTE MYELOID LEUKEMIA
Brief Title: A Study Of PF-06747143, As Single Agent Or In Combination With Standard Chemotherapy In Adult Patients With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to a change in sponsor prioritization.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: B7861002
Record Dates: First submitted 2016-09-21; First posted 2016-11-03 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: relapsed; refractory; acute myeloid leukemia; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Cytarabine; Daunorubicin; Azacitidine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose Escalation (Experimental): Single agent PF-06747143 dose escalation
  Interventions: Biological: PF-06747143
- Cohort 1 (Active Comparator): PF-06747143 with standard dose cytarabine and daunorubicin.
  Interventions: Biological: PF-06747143; Drug: Cytarabine; Drug: Daunorubicin
- Cohort 2 (Active Comparator): PF-06747143 in combination with Azacitidine or Decitabine.
  Interventions: Biological: PF-06747143; Drug: Azacitidine; Drug: Decitabine
- Cohort 3 (Experimental): PF-06747143 dose expansion as a single agent.
  Interventions: Biological: PF-06747143

INTERVENTIONS:
Biological: PF-06747143 — PF 06747143 is a humanized IgG1 monoclonal antibody (mAb) that is an antagonist of CXCR4.
Drug: Cytarabine — 100-200 mg/m2 continuous infusion for 7 days)
  Arms: Cohort 1
Drug: Daunorubicin — 60-90 mg/m2 daily for 3 days
  Arms: Cohort 1
Drug: Azacitidine — 75 mg/m2 sub-cutaneous or intravenous for 7 days)
  Arms: Cohort 2
Drug: Decitabine — 20 mg/m2 continuous intravenous infusion for 5 days in a 4-week schedule
  Arms: Cohort 2

SUMMARY:
Two part, dose escalation and dose expansion study. Open label, multi center, non randomized, multiple dose, safety, pharmacokinetic and pharmacodynamic study of single agent PF-06747143 in sequential dose levels of adult patients with refractory or relapsed AML in order to establish maximum tolerated dose (MTD), recommended Phase 2 dose (RP2D) or maximally permitted dose (MPD) following by a 3 arm dose expansion with PF-06747143 in combination with standard of care chemotherapy in adult patients with AML.

DETAILED DESCRIPTION:
Patients will receive intravenous (IV) PF-06747143 as a weekly infusion (QW) in 28 day cycles at escalating doses. The proposed dosing scheme includes 0.3, 1.0, 3.0, 10, 15, and 20 mg/kg. Patients will be monitored for dose limiting toxicity (DLT) in the dose escalation in order to define the MTD. Two of the three arms in the dose expansion will include PF-06747143 in combination with standard of care chemotherapy and will include a safety lead in. The third arm, pending clinical data, will be PF-06747143 as a single agent.

ELIGIBILITY:
Inclusion Criteria:

Part 1 and Part 2 cohort 3: Patients diagnosed with AML ( bone marrow (BM) or peripheral blood (PB) blast counts >/= 20%) and have received prior chemotherapy and/or standard of care and have relapsed, refractory or Minimal Residual Disease (defined as patients showing residual blast 10-14 days post-induction chemotherapy).

• Patients that are not candidates to receive standard of care and/or refusing the standard care of therapies will also be considered.

Part 2 - Cohort 1 and 2: Newly diagnosed, previously untreated de novo or secondary AML population (AML with bone marrow or peripheral blast counts 20%):

* Cohort 1: Fit to receive intensive remission induction chemotherapy.
* Cohort 2: Unfit to receive or not considered a candidate for intensive remission induction chemotherapy.

Part 1 and 2:

* Life expectancy at least 12 weeks.
* Hydroxyurea is allowed on study to control total peripheral white blood cell count but must be ceased 24 hours prior to first dose.
* Off of prior therapy for 2-4 weeks prior to first dose.
* ECOG performance status: 0 to 2.
* Resolved acute effects of any prior therapy.
* Adequate renal and hepatic function.

Exclusion Criteria:

* Patients with acute promyelocytic leukemia, AML with known central nervous system (CNS) involvement unless the patient has completed treatment for the CNS disease, has recovered from the acute effects of therapy prior to study entry, and is neurologically stable.
* Patient is known refractory to platelet or packed red cell transfusions per institutional guidelines.
* Prior treatment with a compound targeting CXCR4.
* Chronic systemic corticosteroid treatment.
* Known or suspected hypersensitivity to recombinant human proteins.
* Chronic graft versus host disease (GVHD), active GVHD with other than Grade 1 skin involvement, or GVHD requiring systemic immunosuppressive treatment (Part 1 and cohort 3).
* Not recovered from stem cell transplant associated toxicities (Part 1 and cohort 3).
* Prior treatment with hypomethylating agents or chemotherapy for antecedent myelodysplastic syndrome (MDS) (Part 2, cohort 2)
* AML associated with favorable risk karyotypes, including inv(16), t(8;21), t(16;16), or t(15;17) (cohort 2)
* Candidates for allogeneic stem cell transplant (Part 2, cohort 2)
* Known hypersensitivity to cytarabine or daunorubicin (Part 2, cohort 1) and decitabine or azacitidine or mannitol (Part 2, cohort 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2017-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - The University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Banner-University Medical Center Tucson, Tucson, Arizona
  - The University of Chicago Medical Center, Chicago, Illinois
  - Wake Forest Baptist Health, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Liu SH, Gu Y, Pascual B, Yan Z, Hallin M, Zhang C, Fan C, Wang W, Lam J, Spilker ME, Yafawi R, Blasi E, Simmons B, Huser N, Ho WH, Lindquist K, Tran TT, Kudaravalli J, Ma JT, Jimenez G, Barman I, Brown C, Chin SM, Costa MJ, Shelton D, Smeal T, Fantin VR, Pernasetti F. A novel CXCR4 antagonist IgG1 antibody (PF-06747143) for the treatment of hematologic malignancies. Blood Adv. 2017 Jun 21;1(15):1088-1100. doi: 10.1182/bloodadvances.2016003921. eCollection 2017 Jun 27. PMID 29296751
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7861002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to early termination of the study, the planned higher PF-06747143 dose levels (3, 10, 15, and 20 milligrams per kilogram [mg/kg]) in Part 1 were not tested; Part 2 was not conducted.
Groups:
- Part 1: PF-06747143 0.3 mg/kg: PF-06747143 was administered as an intravenous infusion once weekly at 0.3 mg/kg in 28-day cycles.
- Part 1: PF-06747143 1 mg/kg: PF-06747143 was administered as an intravenous infusion once weekly at 1 mg/kg in 28-day cycles.
- Part 1: PF-06747143 at 3 mg/kg: This arm was not initiated due to early termination of the study. PF-06747143 was planned to be administered as an intravenous infusion once weekly at 3 mg/kg in 28-day cycles.
- Part 1: PF-06747143 at 10 mg/kg: This arm was not initiated due to early termination of the study. PF-06747143 was planned to be administered as an intravenous infusion once weekly at 10 mg/kg in 28-day cycles.
- Part 1: PF-06747143 at 15 mg/kg: This arm was not initiated due to early termination of the study. PF-06747143 was planned to be administered as an intravenous infusion once weekly at 15 mg/kg in 28-day cycles.
- Part 1: PF-06747143 at 20 mg/kg: This arm was not initiated due to early termination of the study. PF-06747143 was planned to be administered as an intravenous infusion once weekly at 20 mg/kg in 28-day cycles.
- Part 2: PF-06747143 at MTD/RP2D: This arm was not initiated due to early termination of the study. PF-06747143 at Maximum Tolerated Dose (MTD) or Recommended Phase 2 Dose (RP2D) as an intravenous infusion once weekly in 28-day cycles was optional for Part 2 and planned to be initiated in Part 2 based on single agent PF-06747143 clinical benefit in Part 1.
- Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin: This arm was not initiated due to early termination of the study. PF-06747143 was planned to be administered as an intravenous infusion once weekly at 10 mg/kg in 28-day cycles in combination with standard intensive 7+3 chemotherapy with cytarabine (100-200 mg/m2 continuous infusion for 7 days) and daunorubicin (60-90 mg/m2 daily for 3 days) in Part 2.
- Part 2: PF-06747143 Combined With Azacitidine or Decitabine: This arm was not initiated due to early termination of the study. PF-06747143 was planned to be administered as an intravenous infusion once weekly at 10 mg/kg in 28-day cycles in combination with standard dose of azacitidine (75 mg/m2 administered subcutaneously or intravenously daily for 7 days) or decitabine (20 mg/m2 by continuous intravenous infusion over 1 hour daily for 5 days in a 4-week schedule) in Part 2.
Period: Overall Study
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Part 1: PF-06747143 at 3 mg/kg | Part 1: PF-06747143 at 10 mg/kg | Part 1: PF-06747143 at 15 mg/kg | Part 1: PF-06747143 at 20 mg/kg | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Started | 4 | 4 | 0 (No participants were enrolled in this arm.) | 0 (No participants were enrolled in this arm.) | 0 (No participants were enrolled in this arm.) | 0 (No participants were enrolled in this arm.) | 0 (No participants were enrolled in this arm.) | 0 (No participants were enrolled in this arm.) | 0 (No participants were enrolled in this arm.)
Received Treatment | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but did not receive treatment | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Started another anti-cancer therapy | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Treatment failure and consent withdrawal | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Included all enrolled participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (4) | 63.8 (14.4) | 64.4 (10.5)
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 0 | 1 | 1
  45-64 years | 2 | 0 | 2
  Greater than or equal to (>=) 65 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs) [Part 1]
Description: DLTs were classified according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03 and were defined as any of a predefined set of unacceptable hematologic and non-hematologic adverse events (AEs) occurring in the first treatment cycle unless clearly determined unrelated to PF-06747143. In addition, clinically important or persistent toxicities that were not included in the pre-specified criteria could be considered a DLT following review by the investigators and sponsor.
Time Frame: Day 1 to Day 28 of Cycle 1
Population: All enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg
Number analyzed (Participants) | 3 | 4
Participants | 0 | 1

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) [Part 2]
Description: An AE was any untoward medical occurrence in a participant administered a product or medical device without regard to possibility of causal relationship. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study treatment.
Time Frame: 1 year
Population: No data to report as Part 2 was not conducted.
Arm/Group | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Laboratory Abnormalities [Part 2]
Description: Following parameters were to be analyzed for laboratory examination: hematology (hemoglobin, platelets, white blood cell [WBC], absolute neutrophils, absolute lymphocytes, absolute monocytes, absolute eosinophils, absolute basophils, percent blast cells); chemistry (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase, sodium, potassium, magnesium, chloride, total calcium, total bilirubin, blood urea nitrogen or urea, creatinine, uric acid, glucose [non-fasted], albumin, phosphorous or phosphate); coagulation (prothrombin time [PT] or international normalized ratio [INR], partial thromboplastin time [PTT] or activated PTT [aPTT]); urinalysis (urine dipstick for urine protein: if positive collect 24 hours and microscopic [reflex testing]; urine dipstick for urine blood: if positive collect a microscopic [reflex testing]); pregnancy test (for female participants of childbearing potential, serum or urine).
Time Frame: 1 year
Population: No data to report as Part 2 was not conducted.
Arm/Group | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Objective Response Rate (ORR) - Percentage of Participants With Objective Response [Part 2]
Description: Objective Response was defined as morphologic leukemia-free state (MLFS), complete remission (CR), cytogenetic CR (CRc), molecular CR (CRm), partial remission (PR), or CR or PR with incomplete blood count recovery (CRi or PRi).
  MLFS: Bone marrow (BM) blasts <5%; absence of blasts with Auer rods and extramedullary disease (EMD).
  CR: MLFS criteria; absolute neutrophil count (ANC)>1000/ul and platelet >100,000/ul; independence from red cell transfusions.
  CRc: Reversion to a normal karyotype at the time of CR in cases with an abnormal karyotype at the time of diagnosis; based on the evaluation of 20 metaphase cells from BM.
  CRm: Reversion to a molecular-negative phenotype at the time of CR. CRi: All CR criteria except for ANC <1000/ul or platelet <100,000/ul. PR: ANC >1000/ul and platelet >100,000/ul; BM blasts decreased to 5-25% and ≥50% decrease from pre-treatment levels.
  PRi: ANC <1000/ul or platelet <100,000/ul; BM blasts decreased to 5-25% and ≥50% decrease from pre-treatment levels.
Time Frame: 16 weeks
Population: Part 2 was not conducted.
Arm/Group | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) [Part 1]
Description: An AE was any untoward medical occurrence in a participant administered a product or medical device without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study treatment. AEs included non-serious AEs and SAEs. Causality to study treatment was determined by the investigator.
Time Frame: 1 year
Population: All enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg
Number analyzed (Participants) | 3 | 4
Participants
  AE (all causality) | 3 | 4
  AE (treatment related) | 3 | 3
  SAE (all causality) | 1 | 3
  SAE (treatment related) | 0 | 1

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) by Maximum National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE) Grade [Part 1]
Description: An AE was any untoward medical occurrence in a participant administered a product or medical device without regard to possibility of causal relationship. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study treatment. AEs were graded by the investigator according to NCI CTCAE version 4.03 (Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death related to AE). AEs included non-serious AEs and SAEs.
Time Frame: 1 year
Population: All enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg
Number analyzed (Participants) | 3 | 4
Participants
  Grade 1 | 0 | 0
  Grade 2 | 1 | 0
  Grade 3 | 0 | 0
  Grade 4 | 1 | 3
  Grade 5 | 1 | 1

7. Secondary Outcome: Number of Participants With Hematology Laboratory Abnormalities by Type and Maximum National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE) Grade [Part 1]
Description: Hematology laboratory abnormalities included anemia, hemoglobin increased, lymphocyte count increased, lymphopenia, neutrophil count decreased, platelet count decreased, and white blood cell (WBC) decreased. Each laboratory parameter was graded per NCI CTCAE version 4.03.
Time Frame: 1 year
Population: All enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg
Number analyzed (Participants) | 3 | 4
Participants
  Anemia: Grade 0 | 0 | 0
  Anemia: Grade 1 | 0 | 0
  Anemia: Grade 2 | 0 | 1
  Anemia: Grade 3 | 3 | 3
  Anemia: Grade 4 | 0 | 0
  Hemoglobin increased: Grade 0 | 3 | 4
  Hemoglobin increased: Grade 1 | 0 | 0
  Hemoglobin increased: Grade 2 | 0 | 0
  Hemoglobin increased: Grade 3 | 0 | 0
  Hemoglobin increased: Grade 4 | 0 | 0
  Lymphocyte count increased: Grade 0 | 0 | 4
  Lymphocyte count increased: Grade 1 | 0 | 0
  Lymphocyte count increased: Grade 2 | 3 | 0
  Lymphocyte count increased: Grade 3 | 0 | 0
  Lymphocyte count increased: Grade 4 | 0 | 0
  Lymphopenia: Grade 0 | 0 | 0
  Lymphopenia: Grade 1 | 0 | 0
  Lymphopenia: Grade 2 | 0 | 1
  Lymphopenia: Grade 3 | 0 | 1
  Lymphopenia: Grade 4 | 3 | 2
  Neutrophil count decreased: Grade 0 | 0 | 0
  Neutrophil count decreased: Grade 1 | 0 | 0
  Neutrophil count decreased: Grade 2 | 0 | 0
  Neutrophil count decreased: Grade 3 | 0 | 0
  Neutrophil count decreased: Grade 4 | 3 | 4
  Platelet count decreased: Grade 0 | 0 | 0
  Platelet count decreased: Grade 1 | 0 | 0
  Platelet count decreased: Grade 2 | 0 | 0
  Platelet count decreased: Grade 3 | 0 | 0
  Platelet count decreased: Grade 4 | 3 | 4
  WBC decreased: Grade 0 | 1 | 0
  WBC decreased: Grade 1 | 0 | 1
  WBC decreased: Grade 2 | 0 | 1
  WBC decreased: Grade 3 | 1 | 1
  WBC decreased: Grade 4 | 1 | 1

8. Secondary Outcome: Number of Participants With Chemistry Laboratory Abnormalities by Type and Maximum National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE) Grade [Part 1]
Description: Chemistry laboratory abnormalities included alanine aminotransferase (ALT), alkaline phosphatase, aspartate aminotransferase (AST), bilirubin (total), creatinine, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, and hypophosphatemia. Each laboratory parameter was graded per NCI CTCAE version 4.03.
Time Frame: 1 year
Population: All enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg
Number analyzed (Participants) | 3 | 4
Participants
  ALT: Grade 0 | 0 | 3
  ALT: Grade 1 | 3 | 1
  ALT: Grade 2 | 0 | 0
  ALT: Grade 3 | 0 | 0
  ALT: Grade 4 | 0 | 0
  Alkaline phosphatase: Grade 0 | 0 | 4
  Alkaline phosphatase: Grade 1 | 1 | 0
  Alkaline phosphatase: Grade 2 | 2 | 0
  Alkaline phosphatase: Grade 3 | 0 | 0
  Alkaline phosphatase: Grade 4 | 0 | 0
  AST: Grade 0 | 0 | 1
  AST: Grade 1 | 2 | 3
  AST: Grade 2 | 0 | 0
  AST: Grade 3 | 1 | 0
  AST: Grade 4 | 0 | 0
  Bilirubin (total): Grade 0 | 1 | 2
  Bilirubin (total): Grade 1 | 0 | 1
  Bilirubin (total): Grade 2 | 1 | 1
  Bilirubin (total): Grade 3 | 0 | 0
  Bilirubin (total): Grade 4 | 1 | 0
  Creatinine: Grade 0 | 1 | 2
  Creatinine: Grade 1 | 1 | 1
  Creatinine: Grade 2 | 1 | 1
  Creatinine: Grade 3 | 0 | 0
  Creatinine: Grade 4 | 0 | 0
  Hypercalcemia: Grade 0 | 3 | 4
  Hypercalcemia: Grade 1 | 0 | 0
  Hypercalcemia: Grade 2 | 0 | 0
  Hypercalcemia: Grade 3 | 0 | 0
  Hypercalcemia: Grade 4 | 0 | 0
  Hyperglycemia: Grade 0 | 0 | 1
  Hyperglycemia: Grade 1 | 1 | 2
  Hyperglycemia: Grade 2 | 1 | 1
  Hyperglycemia: Grade 3 | 1 | 0
  Hyperglycemia: Grade 4 | 0 | 0
  Hyperkalemia: Grade 0 | 2 | 3
  Hyperkalemia: Grade 1 | 0 | 1
  Hyperkalemia: Grade 2 | 0 | 0
  Hyperkalemia: Grade 3 | 1 | 0
  Hyperkalemia: Grade 4 | 0 | 0
  Hypermagnesemia: Grade 0 | 2 | 4
  Hypermagnesemia: Grade 1 | 1 | 0
  Hypermagnesemia: Grade 2 | 0 | 0
  Hypermagnesemia: Grade 3 | 0 | 0
  Hypermagnesemia: Grade 4 | 0 | 0
  Hypernatremia: Grade 0 | 3 | 4
  Hypernatremia: Grade 1 | 0 | 0
  Hypernatremia: Grade 2 | 0 | 0
  Hypernatremia: Grade 3 | 0 | 0
  Hypernatremia: Grade 4 | 0 | 0
  Hypoalbuminemia: Grade 0 | 0 | 1
  Hypoalbuminemia: Grade 1 | 0 | 1
  Hypoalbuminemia: Grade 2 | 2 | 2
  Hypoalbuminemia: Grade 3 | 1 | 0
  Hypoalbuminemia: Grade 4 | 0 | 0
  Hypocalcemia: Grade 0 | 0 | 2
  Hypocalcemia: Grade 1 | 1 | 1
  Hypocalcemia: Grade 2 | 1 | 1
  Hypocalcemia: Grade 3 | 1 | 0
  Hypocalcemia: Grade 4 | 0 | 0
  Hypoglycemia: Grade 0 | 3 | 4
  Hypoglycemia: Grade 1 | 0 | 0
  Hypoglycemia: Grade 2 | 0 | 0
  Hypoglycemia: Grade 3 | 0 | 0
  Hypoglycemia: Grade 4 | 0 | 0
  Hypokalemia: Grade 0 | 1 | 1
  Hypokalemia: Grade 1 | 1 | 1
  Hypokalemia: Grade 2 | 0 | 0
  Hypokalemia: Grade 3 | 1 | 2
  Hypokalemia: Grade 4 | 0 | 0
  Hypomagnesemia: Grade 0 | 1 | 1
  Hypomagnesemia: Grade 1 | 2 | 3
  Hypomagnesemia: Grade 2 | 0 | 0
  Hypomagnesemia: Grade 3 | 0 | 0
  Hypomagnesemia: Grade 4 | 0 | 0
  Hyponatremia: Grade 0 | 0 | 2
  Hyponatremia: Grade 1 | 2 | 2
  Hyponatremia: Grade 2 | 0 | 0
  Hyponatremia: Grade 3 | 1 | 0
  Hyponatremia: Grade 4 | 0 | 0
  Hypophosphatemia: Grade 0 | 2 | 2
  Hypophosphatemia: Grade 1 | 0 | 0
  Hypophosphatemia: Grade 2 | 0 | 0
  Hypophosphatemia: Grade 3 | 1 | 2
  Hypophosphatemia: Grade 4 | 0 | 0

9. Secondary Outcome: Objective Response Rate (ORR) - Percentage of Participants With Objective Response [Part 1]
Description: as for outcome 4
Time Frame: 16 weeks
Population: All enrolled participants who received at least 1 dose of study treatment and had a baseline disease assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg
Number analyzed (Participants) | 3 | 4
percentage of participants | NA — Data could not be analyzed as there were 2 treatment failures and 1 non-evaluable participant in this arm. Non-evaluable was due to no post-dose assessment for response. | NA — Data could not be analyzed as there were 2 treatment failures and 2 non-evaluable participants in this arm. Non-evaluable was due to no post-dose assessment for response.

10. Secondary Outcome: Duration of Objective Response Rate (ORR) [Part 1]
Description: Duration of ORR is the time from first documentation of MLFS, CR, CRc, CRm, PR, CRi or PRi to date of first documentation of disease progression or death due to any cause.
  MLFS: BM blasts <5%; absence of blasts with Auer rods and EMD. CR: MLFS criteria; ANC>1000/ul and platelet >100,000/ul; independence from red cell transfusions.
  CRc: Reversion to a normal karyotype at the time of CR in cases with an abnormal karyotype at the time of diagnosis; based on the evaluation of 20 metaphase cells from BM.
  CRm: Reversion to a molecular-negative phenotype at the time of CR. CRi: All CR criteria except for ANC <1000/ul or platelet <100,000/ul. PR: ANC >1000/ul and platelet >100,000/ul; BM blasts decreased to 5-25% and ≥50% decrease from pre-treatment levels.
  PRi: ANC <1000/ul or platelet <100,000/ul; BM blasts decreased to 5-25% and ≥50% decrease from pre-treatment levels.
  Disease progression/relapse: BM blast ≥5%; or reappearance of blast in the blood; or development of EMD.
Time Frame: 16 weeks
Population: All enrolled participants who received at least 1 dose of study treatment and had a baseline disease assessment.
Measure: Median (Full Range); unit: months
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg
Number analyzed (Participants) | 3 | 4
months | NA [NA to NA] — Data could not be analyzed as there were 2 treatment failures and 1 non-evaluable participant in this arm. Non-evaluable was due to no post-dose assessment for response. | NA [NA to NA] — Data could not be analyzed as there were 2 treatment failures and 2 non-evaluable participants in this arm. Non-evaluable was due to no post-dose assessment for response.

11. Secondary Outcome: Progression Free Survival [Part 1]
Description: Progression/relapse free survival is the time from the start of study treatment to first documentation of disease progression or to death due to any cause, whichever occurrs first. Disease progression/relapse: Bone marrow blast ≥ 5%; or reappearance of blast in the blood; or development of extramedullary disease (EMD).
Time Frame: 16 weeks
Population: All enrolled participants who received at least 1 dose of study treatment and had a baseline disease assessment.
Measure: Median (Full Range); unit: months
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg
Number analyzed (Participants) | 3 | 4
months | NA [NA to NA] — Data could not be analyzed as there were 2 treatment failures and 1 non-evaluable participant in this arm. Non-evaluable was due to no post-dose assessment for response. | NA [NA to NA] — Data could not be analyzed as there were 2 treatment failures and 2 non-evaluable participants in this arm. Non-evaluable was due to no post-dose assessment for response.

12. Secondary Outcome: Incidence of Anti-Drug Antibodies (ADA) Against PF-06747143 [Part 1]
Description: Samples were tested for ADA using a validated assay. Number of participants with positive ADA samples was determined.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1, end of treatment
Population: All enrolled patients who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg
Number analyzed (Participants) | 3 | 4
Participants
  Cycle 1 Day 1 | 0 | 1
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 3
  Cycle 1 Day 15 | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 1
  Cycle 2 Day 1 | 0 | 0
  End of treatment | 0 | 0

13. Secondary Outcome: Incidence of Neutralizing Antibodies (Nab) Against PF-06747143 [Part 1]
Description: Samples tested positive for ADA were to be further analyzed for Nab using a validated assay.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1, end of treatment
Population: No data was collected as Nab analysis was not performed.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Incidence of Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (Nab) Against PF-06747143 [Part 2]
Description: Samples were to be analyzed for ADA using a validated assay. ADA positive samples were to be further analyzed for Nab using a validated assay.
Time Frame: Days 1 and 15 pre-dose of Cycle 1, Day 1 pre-dose of Cycles 2-6, Day 1 pre-dose of every 3 cycles thereafter, and at end of treatment
Population: Part 2 was not conducted.
Arm/Group | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of PF-06747143 [Parts 1 and 2]
Description: Cmax of PF-06747143 was the peak serum concentration to be observed directly from data.
Time Frame: Cycle 1 Day 1 at 0, 1, 24, 48, 96 hours; Cycle 1 Day 8 at 0 hour; Cycle 1 Day 15 at 0 and 1 hour; Cycle 1 Day 22 at 0 hour; Cycle 2 Day 1 at 0, 1, 24, 48, 96 hours; Cycle 2 Days 8, 15 and 22 at 0 hour; Subsequent cycles: Day 1 at 0 hour; End of treatment
Population: Due to the early termination of the study, Part 1 pharmacokinetics (PK) assessments were not completed and Part 2 was not conducted.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of PF-06747143 [Parts 1 and 2]
Description: Tmax of PF-06747143 was to be observed directly from data as time of first occurrence of peak serum concentration.
Time Frame: as for outcome 15
Population: Due to the early termination of the study, Part 1 PK assessments were not completed and Part 2 was not conducted.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-06747143 [Parts 1 and 2]
Description: AUClast is area under the serum concentration versus time profile from time zero to the time of the last quantifiable concentration.
Time Frame: as for outcome 15
Population: Due to the early termination of the study, Part 1 PK assessments were not completed and Part 2 was not conducted.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Area Under the Curve From Time Zero to Infinity (AUCinf) of PF-06747143 [Parts 1 and 2]
Description: AUCinf is area under the serum concentration versus time profile from time zero extrapolated to infinite time. If data permitted, AUCinf was to be estimated.
Time Frame: as for outcome 15
Population: Due to the early termination of the study, Part 1 PK assessments were not completed and Part 2 was not conducted.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Apparent Volume of Distribution (Vd) of PF-06747143 [Parts 1 and 2]
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Time Frame: as for outcome 15
Population: Due to the early termination of the study, Part 1 PK assessments were not completed and Part 2 was not conducted.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of PF-06747143 [Parts 1 and 2]
Description: t1/2 is the time measured for the serum concentration to decrease by one half. If data permitted, t1/2 was to be estimated.
Time Frame: as for outcome 15
Population: Due to the early termination of the study, Part 1 PK assessments were not completed and Part 2 was not conducted.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Clearance (CL) of PF-06747143 [Parts 1 and 2]
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 15
Population: Due to the early termination of the study, Part 1 PK assessments were not completed and Part 2 was not conducted.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Maximum Serum Concentration at Steady State (Cmax,ss) of PF-06747143 [Parts 1 and 2]
Description: Assuming steady state was achieved, Cmax,ss was to be determined following multiple dosing to characterize the PK.
Time Frame: as for outcome 15
Population: Due to the early termination of the study, Part 1 PK assessments were not completed and Part 2 was not conducted.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Minimum Observed Serum Trough Concentration at Steady State (Cmin,ss) of PF-06747143 [Parts 1 and 2]
Description: Cmin is the minimum observed serum concentration. Assuming steady state was achieved, Cmin,ss was to be determined following multiple dosing to characterize the PK.
Time Frame: as for outcome 15
Population: Due to the early termination of the study, Part 1 PK assessments were not completed and Part 2 was not conducted.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval at Steady State (AUCtau,ss) of PF-06747143 [Parts 1 and 2]
Description: AUCtau is area under the serum concentration versus time profile from time zero to the time tau (ie, dosing interval). Assuming steady state was achieved, AUCtau,ss was to be determined following multiple dosing to characterize the PK.
Time Frame: as for outcome 15
Population: Due to the early termination of the study, Part 1 PK assessments were not completed and Part 2 was not conducted.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Accumulation Ratio (Rac) of PF-06747143 [Parts 1 and 2]
Description: Accumulation ratio (Rac) was to be obtained from AUCtau at steady state (AUCtau,ss) divided by AUCtau after single dose.
Time Frame: as for outcome 15
Population: Due to the early termination of the study, Part 1 PK assessments were not completed and Part 2 was not conducted.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Clearance (CL) at Steady State of PF-06747143 [Parts 1 and 2]
Description: If data permitted, CL was to be determined following multiple dosing to characterize the PK.
Time Frame: as for outcome 15
Population: Due to the early termination of the study, Part 1 PK assessments were not completed and Part 2 was not conducted.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Volume of Distribution at Steady State (Vss) at of PF-06747143 [Parts 1 and 2]
Description: Vss is the apparent volume of distribution at steady-state. If data permitted, Vss was to be determined following multiple dosing to characterize the PK.
Time Frame: as for outcome 15
Population: Due to the early termination of the study, Part 1 PK assessments were not completed and Part 2 was not conducted.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Terminal Elimination Half-Life (t1/2) at Steady State of PF-06747143 [Parts 1 and 2]
Description: t1/2 is the time measured for the serum concentration to decrease by one half.
Time Frame: as for outcome 15
Population: Due to the early termination of the study, Part 1 PK assessments were not completed and Part 2 was not conducted.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: Peak and Trough PF-06747143 Concentrations for Selected Doses [Part 2]
Description: Peak and trough PF-06747143 concentrations were to be observed directly from data.
Time Frame: as for outcome 15
Population: Part 2 was not conducted.
Arm/Group | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0

30. Primary Outcome: Duration of Objective Response Rate (ORR) [Part 2]
Description: as for outcome 10
Time Frame: 16 weeks
Population: Part 2 was not conducted.
Arm/Group | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0

31. Primary Outcome: Progression Free Survival [Part 2]
Description: as for outcome 11
Time Frame: 16 weeks
Population: Part 2 was not conducted.
Arm/Group | Part 2: PF-06747143 at MTD/RP2D | Part 2: PF-06747143 Combined With Cytarabine and Daunorubicin | Part 2: PF-06747143 Combined With Azacitidine or Decitabine
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Part 1: PF-06747143 0.3 mg/kg | Part 1: PF-06747143 1 mg/kg
All-Cause Mortality (participants affected / at risk) | 3/3 | 1/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/4
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: PF-06747143 0.3 mg/kg (N=3) | Part 1: PF-06747143 1 mg/kg (N=4)
Pyrexia (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: PF-06747143 0.3 mg/kg (N=3) | Part 1: PF-06747143 1 mg/kg (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 2 | 2
Fatigue (General disorders) | 2 | 1
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 3 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to strategic business reasons and was not due to any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT02954653/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT02954653/SAP_001.pdf